CLINICAL TRIAL: NCT02889549
Title: Effects of Different Doses of Ticagrelor and Standard-dose Clopidogrel on Platelet Aggregation and Endothelial Function in Diabetic Patients With Stable Coronary Artery Disease
Brief Title: Effects of Different Doses of Ticagrelor on Platelet Aggregation and Endothelial Function in Diabetic Patients With Stable Coronary Artery Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCAD-20160901
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- Ticagrelor 22.5 mg (Experimental): Ticagrelor (22.5 mg, twice daily, oral) treatment for 1 month.
  Interventions: Drug: ticagrelor
- Ticagrelor 45 mg (Experimental): Ticagrelor (45 mg, twice daily, oral) treatment for 1 month.
  Interventions: Drug: ticagrelor
- Ticagrelor 90 mg (Experimental): Ticagrelor (90 mg, twice daily, oral) treatment for 1 month.
  Interventions: Drug: ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel (75mg, once daily, oral) treatment for 1 month.
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: ticagrelor — Different doses of ticagrelor (22.5/45/90 mg, twice daily, oral) treatment for 1 month
  Arms: Ticagrelor 22.5 mg; Ticagrelor 45 mg; Ticagrelor 90 mg
Drug: clopidogrel — Standard dose of clopidogrel (75 mg, once daily, oral) treatment for 1 month
  Arms: Clopidogrel

SUMMARY:
Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for ACS patients. However, few East Asian patients have been included in these trials to assess the use of these drugs. In addition, a growing body of data supported that East Asian might have different adverse event profiles (thrombophilia and bleeding) and "therapeutic window" compared with white subjects. But it is still not clear whether a low dose of ticagrelor is superior to clopidogrel in diabetic patients with stable coronary disease.

Recent studies found that antiplatelet drugs might have anti-inflammatory effects and protect endothelial function. ACS patients treated by ticagrelor had a significantly higher increase in levels of circulating progenitor cells compared to those treated by clopidogrel, suggesting a benefit on endothelial regeneration that may participate in the pleiotropic property of the drug. This may prompt the regression of blood vessels and the endothelium stability. But it is not very clear that the effect of low-dose ticagrelor on vascular endothelial function in diabetic patients with stable coronary artery disease.

Therefore, the investigators performed this randomized, single-blind clinical trial to observe the effects of different doses of ticagrelor and standard-dose clopidogrel on platelet aggregation and endothelial function in diabetic patients with stable coronary artery disease.

DETAILED DESCRIPTION:
Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for ACS patients. However, few East Asian patients have been included in these trials to assess the use of these drugs. In addition, a growing body of data supported that East Asian might have different adverse event profiles (thrombophilia and bleeding) and "therapeutic window" compared with white subjects. In Korea and Japan, it has been recently reported that low doses of ticagrelor might have a more potent inhibition of platelet aggregation than clopidogrel (75 mg once daily) in healthy subjects and patients with stable coronary artery disease, respectively. But it is still not clear whether a low dose of ticagrelor is superior to clopidogrel in diabetic patients with stable coronary disease. A recent study on pharmacokinetics and tolerability of ticagrelor has found that maximum plasma concentration and area under the plasma concentration-time curve of ticagrelor (90 mg twice daily) and its active metabolite (AR-C124910XX) tended to be approximately 40% higher in healthy Chinese volunteers compared with Caucasian subjects. This data also suggested that a low dose of ticagrelor might be more appropriate for Chinese patients with coronary heart disease. In view of a large diurnal variation with a single daily dose, a lower dose twice daily may be a better choice for Chinese patients.

Recent studies found that antiplatelet drugs might have anti-inflammatory effects and protect endothelial function. ACS patients treated by ticagrelor had a significantly higher increase in levels of circulating progenitor cells compared to those treated by clopidogrel, suggesting a benefit on endothelial regeneration that may participate in the pleiotropic property of the drug. This may prompt the regression of blood vessels and the endothelium stability. But it is not very clear that the effect of low-dose ticagrelor on vascular endothelial function in diabetic patients with stable coronary artery disease.

Therefore, the investigators performed this randomized, single-blind clinical trial to observe the effects of different doses of ticagrelor and standard-dose clopidogrel on platelet aggregation and endothelial function in diabetic patients with stable coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Stable Coronary Artery Disease (1) stable angina (2) low-risk unstable angina (3) variant angina (4) patients with asymptomatic with appropriate therapy（including percutaneous coronary intervention）
2. Diabetes

Exclusion Criteria:

1. ACS
2. planned use of glycoprotein IIb/IIIa receptor inhibitors, adenosine diphosphate (ADP) receptor antagonists, aspirin or anticoagulant therapy during the study period
3. platelet count <100g/L
4. creatinine clearance rate < 30ml/min
5. diagnosed as respiratory or circulatory instability (cardiac shock, severe congestive heart failure NYHA II-IV or left ventricular ejection fraction < 40%)
6. a history of bleeding tendency
7. ticagrelor or clopidogrel allergies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation | up to 1 month

SECONDARY OUTCOMES:
Endothelial Function | up to 1 month

CONTACTS AND LOCATIONS:
Locations (2):
- VerifyNow, San Diego, California, United States
- Endothelial Function detection by brachial artery ultrasound, Harbin, China